CLINICAL TRIAL: NCT06394791
Title: Evaluation of The Efficacy And Safety of Tislelizumab (PD-1) Monoclonal Antibody + IL-2 Combined With Capox Treatment Following Loop Colostomy Surgery in Left-sided Colorectal Cancer Patients Complicating Acute Obstruction
Brief Title: Evaluation of The Efficacy And Safety of PD-1 + IL-2 Combined With Capox Treatment After Loop Colostomy Surgery in Left-sided Colorectal Cancer Patients Complicating Acute Obstruction
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRSYM20240330
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Left-sided Colorectal Cancer Complicating Acute Obstruction
Keywords: Immunotherapy; IL-2; Acute Obstruction
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Tislelizumab with Interleukin-2+CAPOX
  Interventions: Drug: Tislelizumab + IL-2 Combined with Capox

INTERVENTIONS:
Drug: Tislelizumab + IL-2 Combined with Capox — Tislelizumab + IL-2 Combined with Capox

SUMMARY:
Evaluation of The Efficacy And Safety of Tislelizumab (PD-1) Monoclonal Antibody + IL-2 Combined with Capox Treatment Following Loop Colostomy Surgery in Left-sided Colorectal Cancer Patients Complicating Acute Obstruction

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of tumor-related deaths globally, with approximately 40-50% of CRC patients dying from distant metastasis. Current treatments for CRC primarily include surgery, chemotherapy, and targeted therapy, such as monoclonal antibodies against vascular endothelial growth factor (VEGF) and epidermal growth factor receptor (EGFR). However, due to resistance to chemotherapy and targeted therapy, local recurrence or distant metastasis of the tumor, the overall 5-year survival rate for CRC remains low. Therefore, there is an urgent need to develop new treatment methods to improve the prognosis of patients with advanced CRC. The emergence of immunotherapy, including adoptive cell transfer therapy (ACT) and immune checkpoint blockade (ICB), has provided new avenues for the treatment of advanced CRC. However, most CRC patients have limited responses to immunotherapy. For immune checkpoint inhibitors (ICIs), only a minority (15%) of patients with mismatch repair deficiency or high microsatellite instability (dMMR/MSIH) exhibit significant clinical remission. In contrast, most patients with proficient mismatch repair or microsatellite stability (pMMR/MSS) have almost no response to ICIs. In these populations, low tumor mutation burden (TMB) and insufficient immunogenicity leading to inadequate immune cell infiltration are considered major mechanisms of resistance to immunotherapy. Therefore, how to enhance immune cell infiltration and improve the therapeutic effect of immunotherapy in low-responsive CRC remains a critical issue.

In colorectal cancer, the incidence of tumor-associated intestinal obstruction ranges from 8% to 30%, with most obstructions located in the left colon, sigmoid colon, and upper rectum. The most common treatment is emergency surgery to relieve obstruction as soon as possible. However, the risk of anastomotic fistula and the incidence of complications and mortality are relatively high for emergency surgery with proximal and distal bowel anastomosis. Therefore, these patients usually opt for colostomy + staged surgery treatment (Hartmann's procedure). Additionally, due to unstable vital signs, bowel dilation, and bowel and mesenteric edema, comprehensive lymph node dissection and mesenteric resection are limited, which may adversely affect the prognosis of the patient. In recent years, many studies have reported on "stent combined with staged surgery" as a treatment method for left-sided colon cancer with obstruction, but some views believe that stents have the potential risk of compressing the tumor, causing micro-perforation of the intestinal wall leading to local implantation, and increasing the possibility of tumor cell vascular infiltration. Although the waiting period after stent placement can introduce neoadjuvant therapy, existing evidence has not yet proven that stent combined with chemotherapy can effectively downstage the tumor. However, the delay in surgery caused by preoperative chemotherapy does not pose a risk of tumor progression. Current research indicates that acute intestinal obstruction in malignant tumors of the colon exacerbates the body's stress response, including significant accumulation of inflammatory factors such as TNF-α, IL6 throughout the body. Moreover, from a pathophysiological perspective, acute obstruction of colorectal cancer leads to local tissue edema and enhanced inflammatory response, and the tumor tissue may release tumor antigens due to ischemia and necrosis, further inducing the body's immune response. These potential mechanisms provide theoretical support for preoperative neoadjuvant chemotherapy combined with immunotherapy for these patients.

In immunotherapy, the PD-1 inhibition pathway plays a central role in regulating immune cell exhaustion; however, most colorectal cancer patients have limited response to PD-1 monotherapy, hence combining PD1 with other immune-enhancing drugs is hoped to address the above challenges. Currently, some combination therapies have made progress in animal models and are applied in clinical research. Interleukin-2 (IL-2) is a promising candidate drug, synergizing with PD-1 blockade to exert anti-cancer effects. In our phase I clinical study, Capox combined with PD1+IL2 significantly improved the clinical complete remission rate of neoadjuvant therapy for locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 40 and 75 years;
* ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1;
* Tumor tissue samples obtained and histologically confirmed as colon or rectal adenocarcinoma;
* Adequate hematological, liver, and kidney functions: neutrophil count ≥ 1.5×10^9/L; platelet count ≥ 75×10^9/L; serum total bilirubin ≤ 1.5× upper limit of normal (UNL); aspartate aminotransferase ≤ 2.5× UNL; alanine aminotransferase ≤ 2.5× UNL; serum creatinine ≤ 1.5× UNL.

Exclusion Criteria:

* Metastatic disease (Stage IV);
* Recurrent colorectal cancer;
* Concurrent active bleeding, perforation, or other complex situations that cannot be addressed with emergency colostomy surgery alone;
* Previous systemic anti-cancer treatment for colorectal cancer;
* Coexistence of other non-colorectal cancer malignancies;
* Patients with any active autoimmune diseases, or a history of needing steroids or immunosuppressive drugs;
* Patients with interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia);
* Previous treatment-induced any grade 2 or above toxicity reaction (according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5 classification) that has not subsided (excluding anemia, hair loss, and skin pigmentation);
* Previous treatment with anti-programmed death receptor-1 (PD-1) or its ligand (PD-L1) antibodies, anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) antibodies;
* Pregnant or breastfeeding women;
* Known or tested positive for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
* Known or suspected allergy history to any drugs used in the trial;
* Pregnant or breastfeeding women.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Objective Response Rate (CORR) | 18 weeks
  To assess whether neoadjuvant Tislelizumab (PD-1) monoclonal antibody + Interleukin-2 (IL-2) combined with Capox can achieve tumor downstaging

IPD SHARING:
Plan to Share IPD: No